CLINICAL TRIAL: NCT01497496
Title: Phase II Study of Ofatumumab in Combination With High Dose Methylprednisolone Followed by Ofatumumab and Lenalidomide Consolidative Therapy for the Treatment of Relapsed or Refractory CLL/SLL The HiLOG Trial
Brief Title: Ofatumumab/Methylprednisolone and Ofatumumab/Lenalidomide for Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16631; COMB157AUS08T (Other Grant/Funding Number: Novartis); RV-CLL-PI-0560 (Other Grant/Funding Number: Celgene Corp.)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: leukemia; lymphoma; consolidative therapy; combination regimen; Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma | interventions — Methylprednisolone; Adrenal Cortex Hormones; ofatumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunotherapy (Experimental): Combination regimen consisting of high dose methylprednisolone combined with ofatumumab, followed by consolidative therapy with lenalidomide in combination with ofatumumab.
  Interventions: Drug: High Dose Methylprednisolone (HDMP); Drug: Ofatumumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: High Dose Methylprednisolone (HDMP) — 1000 mg/m^2 on Cycle 1: Day 1, 8, 15, 22; Cycle 2: Day 1, 15; Cycle 3: Day 1, 15
  Other Names: HDMP; corticosteroid
Drug: Ofatumumab — Ofatumumab infusion will be administered immediately after HDMP. 300 mg on Cycle 1 Day 1. 2000 mg on Cycle 1: Day 8, 15, 22; Cycle 2: Day 1, 15; Cycle 3: Day 1, 15; Cycle 6: Day 1; Cycle 8: Day 1; Cycle 10: Day 1: Cycle 12: Day 1
  Other Names: Arzerra®
Drug: Lenalidomide — The lenalidomide treatment will start with cycle 4. 5-10 mg pd Days 1-28 as per Creatinine Clearance (CrCl)
  Other Names: Revlimid®; IMiD® compound

SUMMARY:
The main purpose of this study is to see if the combination of ofatumumab with high dose methylprednisolone followed by additional treatment with ofatumumab and lenalidomide can help people with relapsed or refractory CLL/SLL get rid of their CLL/SLL for a long period of time. Researchers also want to find out if the combination of ofatumumab with methylprednisolone followed by additional treatment with ofatumumab and lenalidomide is safe and tolerable.

DETAILED DESCRIPTION:
This is a phase II, single institution, and non-randomized study of patients with relapsed or refractory CLL/SLL, utilizing a two-stage trial design. The primary endpoint for this trial is the combined complete and partial response rate at 3 months (after the end of cycle 3) to the protocol therapy. Investigators anticipate this trial will have a complete response and partial response (CR+PR) rate of at least 55%.

A two-stage design is employed for this trial. The null/unacceptable CR+PR response rate is ≤35% while the anticipated true response rate to the protocol treatment is at least 55% for each disease cohort. At the first stage, 25 patients will be accrued to the trial. If 9 or fewer of these patients respond, then the trial will be terminated early and the response rate to the protocol treatment will be deemed unacceptable (≤35%). Otherwise, if more than 9 patients respond during the first stage, an additional 31 patients will be enrolled to this trial during stage 2 for a total of 56 patients. If 25 or fewer of these 56 patients respond to the protocol treatment at the end of stage 2, no further investigation of the protocol treatment is considered warranted. On the other hand, if more than 25 patients out of the 56 enrolled patients respond, the protocol treatment will be considered promising. If the true response rate is ≤35%, the probability of ending the trial at stage 1 is 0.63. If, however, the true response rate is at least 55%, then the probability of ending the trial at stage 1 is only 0.04. This two-stage design has an overall alpha level of 0.047 and a power of 0.90.

For the purpose of interim analysis at the end of stage 1, the objective response will be measured by the end of 3 months (or end of cycle 3) from the start of the protocol treatment prior to the initiation of the combination of ofatumumab with lenalidomide. The accrual will not be suspended while waiting for the results of the interim analysis unless the observed objective response rate among those patients whose objective response data are available is below 30%.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Patients must have histologically or cytologically confirmed CD5+/CD20+ B-Cell chronic lymphocytic leukemia or small lymphocytic lymphoma. The diagnosis of CLL is based upon the National Comprehensive Cancer Network (NCCN) guidelines. Any outside pathology slides used as inclusion criteria for the patient will be reviewed at this institution to confirm the diagnosis. The patient must meet all of the following CLL criteria to participate in this study: absolute lymphocyte count > 5000/μL; CD20+ and CD5+; Bone marrow (BM) lymphocytes ≥ 30%; Or previous confirmed diagnosis of CLL/SLL with less than 5000/μl or less than 30% lymphocytes in BM.
* Patients are eligible if they have relapsed or refractory CLL/SLL.
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry
* Laboratory test results within these ranges: Absolute neutrophil count ≥ 1000/mm³, Platelet count ≥50,000 /mm³, Renal function assessed by calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula, Total bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartic transaminase (AST/SGOT) and alanine transaminase (ALT/SGPT) ≤ 2.5 x ULN, Alkaline phosphatase <2.5 x ULN
* Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid (ASA) may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide)
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Evidence of laboratory Tumor Lysis Syndrome (TLS) by Cairo-Bishop Definition. Patients may be enrolled upon correction of electrolyte abnormalities.
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV)
* Positive serology for hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive and HBsAb negative, a HB DNA test will be performed and if positive the patient will be excluded. Note: If HBcAb positive and HBsAb positive, which is indicative of a past infection, the patient can be included. Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Positive serology for hepatitis C (HC) defined as a positive test for hepatitis C antibodies (HCAb), in which case reflexively perform a HC recombinant immunoblot assay (RIBA) on the same sample to confirm the result
* Patients who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment) are ineligible.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to randomization, congestive heart failure [New York Heart Association (NYHA) III-IV], and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-01-26 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Bello, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Immunotherapy: Combination regimen consisting of high dose methylprednisolone combined with ofatumumab, followed by consolidative therapy with lenalidomide in combination with ofatumumab. Time of therapy: until disease progression or toxicity.
Period: Overall Study
Arm/Group | Immunotherapy
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Immunotherapy
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR at 3 months. Assessment for response will be made following the National Cancer Institute Working Group (NCIWG) 2008 Chronic Lymphocytic Leukemia (CLL) criteria for response. Objective response = Complete Response (disappearance of all target lesions) + Partial Response (>=30% decrease in the sum of the longest diameter of target lesions) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0)
Time Frame: 3 Months
Population: Evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Immunotherapy
Number analyzed (Participants) | 27
percentage of participants | 48.3

2. Secondary Outcome: Rate of Progression-free Survival (PFS)
Description: Progression-free survival (PFS), defined as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier, will be summarized with the Kaplan-Meier curve. Progressive Disease (PD) defined according to NCIWG 2008 CLL Criteria for Response.
Time Frame: 36 Months
Population: Data not collected (likely futility from low accrual due to competing commercially available treatment)
Arm/Group | Immunotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Overall Survival (OS)
Description: Overall Survival Time: Time from initiation of treatment to time of death. Overall survival will be summarized with the Kaplan-Meier curve.
Time Frame: 36 Months
Population: Data not collected (likely futility from low accrual due to competing commercially available treatment)
Arm/Group | Immunotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 7 years, 6 months
Arm/Group | Immunotherapy
All-Cause Mortality (participants affected / at risk) | 5/29
Serious Adverse Events (participants affected / at risk) | 25/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy (N=29)
Anemia (Blood and lymphatic system disorders) | 4 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (13)
Leukocytosis (Blood and lymphatic system disorders) | 2 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 1 (1) — C-diff
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1) — bleed from right ear lesion
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 1 (1)
General disorders and administrative site conditions -Other (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 6 (6)
Lung infection (Infections and infestations) | 9 (10)
Sepsis (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 25 (107)
Platelet count decreased (Investigations) | 8 (23)
White blood cell decreased (Investigations) | 12 (36)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Penumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Vascular disorders - Other (Vascular disorders) | 1 (1) — pulmonary embolus
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy (N=29)
Anemia (Blood and lymphatic system disorders) | 6 (8)
Intermittent anemia (Blood and lymphatic system disorders) | 2 (2)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1) — Bleeding tendency
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis -leukopenia (Blood and lymphatic system disorders) | 1 (2)
Intermittent Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain - abdominal (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain - pain & swelling (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) — bigeminy
Cardiac disorders - Other (Cardiac disorders) | 1 (1) — carotid stenosis
Cardiac disorders -other (Cardiac disorders) | 2 (2) — chest tightness
Cardiac disorders - Other (Cardiac disorders) | 1 (1) — hypokinesis inferior wall of left ventricle
Cardiac disorders - Other (Cardiac disorders) | 1 (1) — systolic murmur
Palpitations (Cardiac disorders) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Hearing impairment (Ear and labyrinth disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) — possible ear infection
Vertigo (Ear and labyrinth disorders) | 2 (2)
Endocrine disorders Other (Endocrine disorders) | 1 (1) — Heat intolerance
Endocrine disorders - Other (Endocrine disorders) | 1 (1) — mild dysphonia
Blurred vision (Eye disorders) | 4 (4)
visual disturbances (Eye disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 6 (6)
Eye pain (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (3)
Watering eyes (Eye disorders) | 1 (1)
Abdominal cramping (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (10)
Abdominal bloating (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 17 (21)
Diarrhea (Gastrointestinal disorders) | 16 (31)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal reflux disease (Gastrointestinal disorders) | 5 (11)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 1 (1) — burning sensation mouth
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — diverticulosis
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — hiatal hernia
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — increased belching
Gastrointestinal pain (Gastrointestinal disorders) | 2 (3)
Gastroparesis, mild (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea, intermittent (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 12 (13)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting, intermittent (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9)
Chills (General disorders) | 10 (11)
Rigors (Gastrointestinal disorders) | 2 (2)
Edema, face (General disorders) | 2 (2)
Edema, limbs (General disorders) | 12 (21)
Fatigue (General disorders) | 16 (24)
Fever (General disorders) | 12 (17)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1) — balance problems, intermittent
Gait disturbance (General disorders) | 1 (1) — difficulty walking/coordination
Gait disturbance (General disorders) | 1 (1)
Hemorrhoids (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 4 (4)
Irritability (General disorders) | 6 (6)
Malaise (General disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Left hip pain (General disorders) | 1 (1)
port pain (General disorders) | 1 (1)
throat pain (General disorders) | 1 (1)
Inguinal pain, groin pain (General disorders) | 2 (2)
General disorders - Other (General disorders) | 1 (1) — pain shoulder/mediport catheter
Upper axilla pain (General disorders) | 1 (1)
hip pain (General disorders) | 2 (2)
General disorders - Other (General disorders) | 1 (1) — Arm pain due to fall
Joint pain (General disorders) | 1 (1)
Shooting pain, right leg (General disorders) | 1 (1)
Wrist pain (General disorders) | 1 (1)
Gallbladder polyps (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 5 (5)
Cytokine release syndrome (Immune system disorders) | 3 (3)
Bronchial infection (Infections and infestations) | 2 (2)
Enterocolitis infections (Infections and infestations) | 2 (2)
Infections and Infestations - Other (Infections and infestations) | 4 (5)
Lung infection (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinitis ineffective (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 3 (5)
Upper respiratory infection (Infections and infestations) | 7 (13)
Urinary tract infection (Infections and infestations) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 3 (3)
Papular lesion on face (Injury, poisoning and procedural complications) | 1 (1)
alamine aminotransferase increased (Investigations) | 5 (10)
Alkaline phosphatase increased (Investigations) | 5 (12)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Blood bilirubin increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 5 (7)
Investigations - Other (Investigations) | 5 (5)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 22 (94)
Platelet count decreased (Investigations) | 11 (26)
Weight loss (Investigations) | 4 (5)
White blood cell decreased (Investigations) | 22 (115)
Anorexia (Metabolism and nutrition disorders) | 9 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (34)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 10 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (7)
Muscle weakness, lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 (4) — Muscle aches, spasms
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Neoplasms benign, malignant and unspecified -Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (11)
Akathisia (Nervous system disorders) | 2 (5)
Ataxia (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 10 (15)
Dysgeusia (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 7 (14)
Memory impairment (Nervous system disorders) | 2 (2)
Movement, involuntary (Nervous system disorders) | 9 (10)
Nervous system disorders - Other (Nervous system disorders) | 4 (4)
Parasthesia (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (21)
Tremor (Nervous system disorders) | 7 (7)
Agitation (Psychiatric disorders) | 6 (7)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 13 (13)
Personality change (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 10 (11)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Reespiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 (4)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 (16)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (11)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 11 (16)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Surgical and medical procedures - Other (Surgical and medical procedures) | 4 (9)
Flushing (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (8)
Hypotension (Vascular disorders) | 4 (4)
Vascular disorders - Other (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT01497496/Prot_SAP_000.pdf